CLINICAL TRIAL: NCT06776146
Title: Proteomic Profiling to Differentiate Pancreatic and Biliary Adenocarcinomas
Acronym: PROFIPANC-CHOL
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/94
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; Biliary adenocarcinoma; Diagnosis; Proteomic; Proteomic profiling
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- pancreatic adenocarcinomas: Patients with pancreatic adenocarcinomas
  Interventions: Diagnostic Test: proteomic profiling
- distal cholangiocarcinomas: Patients with distal cholangiocarcinomas
  Interventions: Diagnostic Test: proteomic profiling
- pancreatobiliary adenocarcinomas with diagnostic challenges: Patients with pancreatobiliary adenocarcinomas with diagnostic challenges
  Interventions: Diagnostic Test: proteomic profiling

INTERVENTIONS:
Diagnostic Test: proteomic profiling — proteomic profiling

SUMMARY:
Distal cholangiocarcinoma and pancreatic adenocarcinoma are aggressive cancers with overlapping diagnostic features, making them challenging to differentiate. Although both require similar surgical treatment, their postoperative chemotherapy regimens differ significantly, with capecitabine used for distal cholangiocarcinoma and modified FOLFIRINOX for pancreatic adenocarcinoma, based on distinct guidelines. In 10-20% of cases, due to their close anatomical proximity, pathologists cannot distinguish between these cancers, leading to diagnostic uncertainty and potential therapeutic missteps. Proteomic profiling, a cutting-edge technique leveraging protein analysis for diagnostic precision, could offer a novel solution to this challenge, although it has yet to be applied in this context

DETAILED DESCRIPTION:
Distal cholangiocarcinoma (also known as biliary adenocarcinoma) and pancreatic adenocarcinoma are two aggressive cancers with numerous diagnostic similarities. They often present with nearly identical clinical features, tumor markers, and imaging findings on computed tomography (CT). Both cancers require similar surgical management-namely, a pancreaticoduodenectomy (also known as the Whipple procedure)-but their adjuvant systemic chemotherapy protocols in the postoperative setting differ significantly.

According to the French guidelines from the National Digestive Cancer Thesaurus, patients operated on for distal cholangiocarcinoma receive capecitabine as adjuvant therapy, while those treated for pancreatic adenocarcinoma receive modified FOLFIRINOX. These recommendations are based on randomized prospective studies that demonstrated improved overall survival and recurrence-free survival with these specific therapeutic regimens for each cancer. Thus, selecting the appropriate chemotherapy tailored to the cancer type is crucial for patient outcomes.

However, due to the close anatomical proximity of these two tumors-since the bile duct traverses the pancreatic head-it is estimated that in 10-20% of cases, the pathologist is unable to distinguish between these cancers. In such instances, the diagnosis is reported as "adenocarcinoma of pancreatobiliary origin." This ambiguity forces clinicians to choose a chemotherapy regimen based on a combination of clinical, radiological, and pathological findings rather than definitive histological evidence, thereby increasing the risk of an inappropriate treatment choice.

Proteomic profiling is an innovative analytical technique that enables diagnostic insights by analyzing the complete protein composition of a tissue sample and matching it to predefined profiles using statistical algorithms. While this method has already been successfully employed to aid in the diagnosis of other conditions-such as hepatocellular adenomas, amyloidosis, and biliary strictures of indeterminate origin-it has not yet been applied to differentiate pancreatic adenocarcinoma from distal cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Pancreaticoduodenectomy for pancreatic adenocarcinoma or distal cholangiocarcinoma
* Patient's non-opposition to the reuse of data

Exclusion Criteria:

* Neoadjuvant chemotherapy
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 patients with pancreatic adenocarcinomas, 10 patients with distal cholangiocarcinomas, 8 patients presenting pancreatobiliary adenocarcinomas with diagnostic challenges
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
proteomic signature | baseline
  proteomic signature capable of differentiating cholangiocarcinoma from pancreatic adenocarcinoma through proteomic profiling of surgical specimens

SECONDARY OUTCOMES:
diagnostic biomarkers | baseline
  diagnostic biomarkers applicable in immunohistochemistry to differentiate cholangiocarcinoma from pancreatic adenocarcinoma based on proteomic analyses

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No